CLINICAL TRIAL: NCT03160300
Title: Placebo-Controlled, Randomized, Double-Blind Trial on the Effect of Binaural Beats on Pain Perception and Analgesic Medication Use in Patients Suffering From Chronic Pain
Brief Title: The Effect of Binaural Beats on Pain Perception and Analgesic Medication Use in Patients Suffering From Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vasileios Gkolias, MD, MSc, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Binaural Beats Pain
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binaural Beats (Experimental): Music with Binaural Beats: Binaural beat signals embedded in relaxing music, in a crossover design
  Interventions: Device: Music with Binaural Beats
- Placebo (Sham Comparator): Music: Relaxing music without the binaural beat component, in a crossover design
  Interventions: Device: Music

INTERVENTIONS:
Device: Music with Binaural Beats — Relaxing music with embedded binaural beats at a frequency of 5 Hz
  Arms: Binaural Beats
Device: Music — Relaxing music without a binaural beat component
  Arms: Placebo

SUMMARY:
This study evaluates the effect of binaural beats on pain perception and subsequent need for analgesic medication use in patients suffering from diseases causing chronic pain. All patients will receive two consecutive interventions: binaural beat signals embedded in relaxing music and placebo (relaxing music without the binaural beat component), in random order.

DETAILED DESCRIPTION:
Binaural beats consist of two artificially produced sound waves, differing in wave frequency, presented simultaneously and separately to each ear. The brain, following binaural beat processing, synchronizes to the frequency difference between the two waves. Therefore, using a 5 Hz frequency difference (theta rhythm), which promotes relaxation, we could alleviate pain perception and subsequent analgesic medication use.

Patients suffering from chronic pain will receive two consecutive interventions: binaural beat signals embedded in relaxing music and placebo (relaxing music without the binaural beat component), in random order.

Electroencephalogram (EEG) recordings will be used to confirm brain frequency synchronization, whereas pain severity scales and a diary recording analgesic medication use will be used to identify differences between intervention and placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain
* Regular analgesic medication use

Exclusion Criteria:

* Malignant pain
* Headache as the cause of chronic pain
* Hearing disability
* Neuropsychiatric disease
* Previous experience with binaural beats

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Effect on pain severity | After 30 minutes of listening to binaural beat signals or sham intervention
  Comparing pre- and post-intervention perceived pain levels, using a Numeric Rating Scale (NRS) 0-10
Effect on analgesic medication use | One week on an "as needed" basis intervention use to alleviate pain, keeping a diary
  Comparing analgesic medication active substance quantity used, documented on patient diary recordings

SECONDARY OUTCOMES:
Effect on electroencephalogram (EEG) | 30 minutes of listening to binaural beat signals or sham intervention
  Evaluating differences in post-intervention EEG rhythm, using advanced biomedical signal processing, compared to baseline EEG rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Kouvelas, Professor, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided